CLINICAL TRIAL: NCT07282899
Title: Overview of Intraoperative Lung Protective Ventilation in Czech Republic
Brief Title: Intraoperative Lung Protective Ventilation in Czech Republic
Acronym: IOLPVCZ
Status: Not yet recruiting | Type: Observational
Sponsor: Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s. (Other)
Responsible Party: Principal Investigator, Michal Kalina, deputy for science and research, Masarykova Nemocnice v Usti nad Labem, Krajska Zdravotni a.s.
Other Study IDs: IOLPVCZ
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Intraoperative Lung Protective Ventilation
Keywords: general anaesthesia; intraoperative lung protective ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This questionnaire-based study aims to evaluate the adherence to and current clinical practices regarding intraoperative lung-protective ventilation (IOLPV) among anesthesiologists in the Czech Republic. Despite the established role of IOLPV in reducing postoperative pulmonary complications in selected populations, its routine application during general anesthesia for elective surgeries remains variable. The survey focuses on identifying common ventilation strategies, attitudes toward lung recruitment maneuvers, tidal volume selection, use of PEEP, and awareness of existing recommendations. The results will provide insight into national practice patterns, perceived barriers, and educational needs, helping to inform future guidelines, training initiatives, and efforts to enhance patient safety and postoperative outcomes across Czech anesthesia departments.

DETAILED DESCRIPTION:
This study is designed as an observational cross-sectional survey focusing on attitudes, knowledge, and practical application of intraoperative lung-protective ventilation among anesthesiology professionals in the Czech Republic. The primary aim is to describe the prevalence of LPV-related practices during general anesthesia in adult surgical patients. Key elements of LPV include the use of lower tidal volumes adjusted to predicted body weight, titrated PEEP, avoidance of unnecessary high oxygen fractions, and a judicious approach to lung recruitment maneuvers. The study evaluates whether these components are routinely utilized and if so, under what clinical circumstances.

Secondary aims of the study include identifying barriers that may prevent anesthesiologists from applying LPV techniques, such as concerns about hemodynamic instability, limited training, lack of standardized protocols, insufficient monitoring capabilities, or doubts regarding clinical benefit. The survey also investigates how clinicians perceive the safety of recruitment maneuvers and whether they encounter adverse effects such as hypotension, desaturation, or barotrauma. The survey explores whether respondents view LPV as universally beneficial or applicable only to specific patient groups such as obese or critically ill individuals. The study further investigates whether national or departmental protocols and guidelines for ventilation exist at respondents' workplaces, whether ventilator settings are standardized, and whether institutional education or quality improvement initiatives support evidence-based ventilation.

The target population consists of anesthesiologists and anesthesiology trainees actively involved in perioperative care in hospitals across the Czech Republic. Participation is voluntary and anonymous, with no patient-level data collected. Demographic information such as level of training, years of experience, type of institution, and exposure to specialized perioperative or intensive care practice is included to allow subgroup comparisons. Data collection is conducted online via a secure electronic questionnaire with an estimated completion time of approximately five to eight minutes. The distribution strategy includes professional organizations, departmental mailing lists, and professional association communication channels to maximize nationwide representation.

The study utilizes a structured questionnaire composed of multiple-choice and ordinal-scale items that address five thematic categories: general anesthetic ventilation practices including tidal volume and FiO₂ selection; PEEP use and adherence to recommendations; indications and frequency of recruitment maneuvers; perceived safety and complications associated with LPV; and institutional culture, including guideline availability and ventilator technology. Respondents are asked to report how they usually manage typical elective surgical cases rather than unusual or high-risk scenarios, allowing insight into real-world standard practices. The results will quantify how closely routine clinical practice aligns with currently available scientific evidence and international perioperative ventilation recommendations.

The primary outcome is the proportion of respondents reporting ventilation settings that meet predefined LPV criteria in their routine practice. Secondary outcomes include differences in adherence between trainee and consultant anesthesiologists, between academic and non-academic hospitals, between centers with and without formal local protocols, and between clinicians with differing exposure to intensive care medicine. The data will be analyzed descriptively and comparatively to identify significant trends or variability within the national practice environment. Findings from this survey may provide a basis for future interventional or educational studies and facilitate development of nationwide recommendations.

The study is conducted in accordance with ethical research principles, including the Declaration of Helsinki and relevant European data protection regulations. Ethical approval is being obtained prior to survey initiation. Participation is fully voluntary, and no identifying personal data are collected; responses are recorded and analyzed only in aggregated form. No clinical intervention is performed, and therefore no additional risks to patients or participants are expected. The expected benefits of this research include improved understanding of current perioperative respiratory practices and identification of potential gaps where updated knowledge translation or institutional support may be necessary.

The overall purpose of this project is to contribute to improving perioperative patient outcomes by strengthening evidence-based ventilation strategies during general anesthesia. By highlighting current practice and potential challenges in implementation, the results can support targeted educational efforts, standardized national recommendations, and greater awareness of intraoperative pulmonary protection among Czech anesthesia providers. The data will also help position Czech clinical practice within the broader European context and may encourage future collaborative research initiatives focused on postoperative pulmonary complication reduction and enhanced quality of anesthesia care.

ELIGIBILITY:
Inclusion Criteria:

* anaesthesiologist practiting in Czech republic

Exclusion Criteria:

* not lincensed anaesthesiologist
* anaesthesiologist outside Czech republic

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Anaesthesiologists in Czech republic
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to IOLPV | 20 days
  Number of respondents that respond that meet IOLPV guidelines

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared through research office of the main department of the principal investigator on reasonable request.